CLINICAL TRIAL: NCT03321448
Title: Novel Tumor Targeted Fluorescent TMTP1-ICG Mapping in Laparoscopic Sentinel Lymph Node Detection in Cervical Cancer Patients
Brief Title: TMTP1-ICG Mapping in Laparoscopic SLN Detection in Cervical Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ding Ma, Director, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TMTP1-ICG-01
Record Dates: First submitted 2017-10-23; First posted 2017-10-25 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMTP1 (Experimental): The TMTP1-ICG (WuXi AppTec, Shanghai, China) powder was diluted in 20 ml of aqueous sterile water to a concentration of 1.0 mg/mL. 0.4ml of this TMTP1-ICG solution was injected into the cervix, divided into 3 and 9 o'clock position, in the operating room. During the laparoscopy, the PinPoint S1 Novadaq (PinPoint Endoscopic Fluorescence Imaging System, NOVADAQ, Mississauga, ON, Canada), 30° laparoscopes were used for fluorescent detection.
  Interventions: Drug: TMTP1-ICG
- ICG (Active Comparator): The ICG powder was diluted in 20 ml of aqueous sterile water to a concentration of 1.0 mg/mL. 0.4ml of ICG solution was injected into the cervix, divided into 3 and 9 o'clock position, in the operating room. During the laparoscopy, the PinPoint S1 Novadaq (PinPoint Endoscopic Fluorescence Imaging System, NOVADAQ, Mississauga, ON, Canada), 30° laparoscopes were used for fluorescent detection.
  Interventions: Drug: ICG

INTERVENTIONS:
Drug: TMTP1-ICG — Detection of SLN
  Arms: TMTP1
Drug: ICG — Detection of SLN
  Arms: ICG

SUMMARY:
investigators aimed to determine the validity of our novel tumor targeted fluorescent TMTP1-ICG to increased accuracy of laparoscopic SLN mapping

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, married, without childbearing requirements at the time of consent.
* FIGO stage IA1-IIB cervical squamous cell cancer and is a candidate for laparoscopy intervention, with lymph node dissection being a part of the surgical plan.
* Subject has provided written informed consent.

Exclusion Criteria:

* Breast-feeding or pregnant
* Ongoing participation in another clinical trial with an investigational drug with 3 months
* Own allergy towards ICG and/or alcohol
* Diagnosis of bacterial vaginosis, fungal vaginitis, sexually transmitted diseases
* Patients with cardiac dysfunction or hepatic insufficiency or renal insufficiency

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Detection rate of sentinel lymph node | 1 day
  Detection of sentinel lymph node per patient

SECONDARY OUTCOMES:
Sensitivity | 7 days
  Sensitivity of SLN mapping of TMTP1-ICG compared to the sensitivity of SLN mapping of ICG
Specificity | 7 days
  Specificity of SLN mapping of TMTP1-ICG compared to the sensitivity of SLN mapping of ICG
Incidence of adverse events | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical Colledge, HUST, Wuhan, Hubei, China